CLINICAL TRIAL: NCT06860568
Title: Annotation of Geographic Atrophy in Hyperspectral Images Captured With the Optina-4C™
Brief Title: The GA in HSI Study
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-24-015
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Geographic Atrophy; Healthy
MeSH Terms: conditions — Geographic Atrophy | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Eyes of patients with a diagnosis of dry AMD with GA lesions
  Interventions: Other: Retrospective Study
- Cohort B: Eyes of patients with a diagnosis of AMD without the presence of RPE disruptions
  Interventions: Other: Retrospective Study
- Cohort C: Eyes of age-matched healthy patients (no AMD or GA lesions)
  Interventions: Other: Retrospective Study

INTERVENTIONS:
Other: Retrospective Study — Retrospective Study This study will use a retrospective Test Dataset of eye scans collected by Optina under different study protocols. MHRC H5 Images collected as part of Optina studies CIP-22-003, CIP-22-004, DOC100463 or RWD-24-011 will be reviewed by an Optina Data Analyst and flagged for potential match to the Target Population. Of the flagged images, 40 will be selected and allocated to the Test Dataset. All selected images must have a matching OCT image for review as part of the Reference Data. The Test Dataset will be documented in the CIP-24-015 data spreadsheet and archived in the CIP-24-015 central files.

SUMMARY:
This study used a retrospective dataset collected by Optina under different study protocols. The target study population will include adults over the age of 50 years, with and without the presence of AMD.

DETAILED DESCRIPTION:
This retrospective, case-control study used the clinical data previously collected by Optina (CIP 22-003 AND Study, CIP 22-004 CAS Training Study and RWD 24-011 RWD Study). As such, no new participants were enrolled for this study. The review and annotation of the MHRC H5 Images for GA are within the scope of each of these studies and the study participants have provided their Informed Consent for use of their retinal scans to assess clinical diagnostic applications. Images from the above-mentioned studies that met the inclusion criteria (there were no exclusion criteria) were classified into 3 different cohorts per the selection process described in the Study Protocol. Each cohort required a minimum of 10 MHRC Images from unique eyes with matched OCT scans.

* Cohort A: Eyes of patients with a diagnosis of dry AMD with GA lesions:

  o This cohort included patients with intermediate-or late-stage dry AMD where GA lesions are present, based on either the diagnostic information provided by the clinic, or by visible assessment of either the HSI or OCT images performed by the Optina Analyst.
* Cohort B: Eyes of patients with diagnosis of dry AMD without the presence of GA lesions

  o This cohort included patients with early or intermediate dry AMD where GA lesions are not present, based on either the diagnostic information provided by the clinic, or by visible assessment of either the HSI or OCT images performed by the Optina Analyst.
* Cohort C: Eyes of age-matched healthy patients (no AMD or GA lesions)

  * This cohort included patients with healthy retinas, based on either the diagnostic information provided by the clinic, or by visible assessment of either the HSI or OCT images performed by the Optina Analyst. Knowledge Transfer and Training Optina facilitated a Knowledge Transfer and Training session by the IOI for CapeStart Study Personnel.

CapeStart Study Personnel were trained in using Optivizon Viewing Software, the viewing software included in the marketed version of Optina-4C (MHRC device), and the Optina Segmentation tool.

Additionally, they were trained in the presentation of GA in HSI Images. Evaluation Phase CapeStart were provided with the Test Dataset of eye scans (n=40 eyes). CapeStart Optometristsreviewed all the HSI Images from the Optina-4C in Optivizon, annotated any GA lesions (if present) in the RelSpec@560 image using the Optina Segmentation tool, and completed the HSI Questionnaire for the MHRC H5 Images. Annotation Process The HSI RelSpec@560 Images were annotated by the CapeStart Optometrists for the Evaluation Phase.

The annotations were completed using the validated Optina Segmentation Tool per the User Manual, and all image annotations were performed on the Virtual Machine established and validated by Optina for this study.

If the eye was considered to have at least one GA lesion after viewing the MHRC H5 Images in Optivizon, the RelSpec@560 Image was annotated using the Optina Segmentation Tool. The annotator used the yellow label for high confidence level for GA visualization and Blue label for low confidence level.

Reference Data The IOI was responsible for generating the reference data. The IOI reviewed all OCT images as well as the MHRC H5 Images, then annotated the RelSpec@560 images. The IOI visual assessment made note of all cRORA (GA lesions) and iRORA (nascent GA lesion) in the OCT and aligned where possible with corresponding lesions in the HSI images. Lastly, the IOI completed the HSI Questionnaire for all annotated Relspec images.

ELIGIBILITY:
Inclusion Criteria:

Participants may enter the study only if ALL the following inclusion criteria are present:

* Study participants over the age of 50 years who consented to participate in Optina studies CIP-22-003, CIP-22-004, DOC100463, or RWD-24-011.
* MHRC H5 Image Cube has been reviewed by an Optina Analyst and identified as aligned with the Target Population (see Section 5.2).
* MHRC H5 Image Cube has a corresponding OCT image.

Exclusion Criteria:

* No exclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will use a retrospective dataset collected by Optina under different study protocols. The target study population will include adults over the age of 50 years, with and without the presence of AMD.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Comparison of the total number of Relspec images annotated for GA lesions | 45 days
  Comparison of the total number of Relspec images annotated for GA lesions of at least 29 pixels or larger with the total number of OCT images with identified GA lesions (cRORA) in the Test Dataset.
Comparison of the total number of 'high certainty' GA lesions | 45 days
  Comparison of the total number of 'high certainty' GA lesions (Yellow label) of at least 29 pixels annotated in all Relspec images with the total number of (cRORA) identified in the OCT images in the Test Dataset.
Comparison of the total number of GA lesions | 45 days
  Comparison of the total number of GA lesions (Yellow label and Dark Blue label) of at least 29 pixels or larger annotated in all Relspec images with the total number of identified GA lesions (cRORA) in the OCT images in the Test Dataset.
Evaluation of the Global DICE Score | 45 days
  Evaluation of the Global DICE Score for annotations of 29 pixels or larger performed by CapeStart compared with the Reference Data.

CONTACTS AND LOCATIONS:
Overall Officials: Ramina Nissan, OD, Principal Investigator — The Glen Site, McGill University Health Centre
Locations (1):
- Optina Diagnostics Inc, Montreal, Quebec, Canada